CLINICAL TRIAL: NCT00298415
Title: Phase III Study of Monotherapy by Gemcitabine or Vinorelbine Comparing to Doublet by Carboplatin and Paclitaxel Among Elderly Patients With Stage IIIB/IV NSCLC (Obligatory Second-line by Erlotinib)
Brief Title: Chemotherapy of Elderly Patients With Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFCT-0501
Record Dates: First submitted 2006-03-01; First posted 2006-03-02 (Estimated); Last update posted 2013-10-25 (Estimated); Status verified 2013-10

CONDITIONS: NSCLC
Keywords: 2-years survival
MeSH Terms: interventions — CP protocol; Gemcitabine; Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Chemotherapy (mono)
  Interventions: Drug: Monotherapy (gemcitabine or vinorelbine)
- B (Experimental): Chemotherapy (doublet)
  Interventions: Drug: Paclitaxel + Carboplatin

INTERVENTIONS:
Drug: Paclitaxel + Carboplatin — Paclitaxel 90 mg/m² D1, D8, D15 (D1=D29, 4 cycles) Carboplatin AUC 6 D1 (D1=D29, 4 cycles)
  Other Names: Treatment after progression : Erlotinib 150 mg/day
  Arms: B
Drug: Monotherapy (gemcitabine or vinorelbine) — Gemcitabine 1150 mg/m² D1 and D8 (D1=D22, 5 cycles) Vinorelbine 30 mg/m² D1 and D8 (D1=22, 5 cycles)
  Other Names: Treatment after progression : Erlotinib 150mg/day
  Arms: A

SUMMARY:
The last ASCO recommendations in 2003 for the treatment of a CBNPC of stage IIIB/IV of elderly people, are to manage a monochemotherapy. Paclitaxel in association with carboplatin is feasible in elderly patients and the retrospective analysis of two studies of the comparing SWOG, one this association with that of cisplatine and vinorelbine and the other cisplatine only with cisplatine and vinorelbine, showed among 117 the 70 years old patients and more, the absence of significant difference of survival and toxicity compared to the younger patients. The study recently published of Lilenbaum and Al shows that among patients with bad PS, association carboplatine and paclitaxel do better than the paclitaxel only. The paclitaxel managed in weekly form is likely of a better activity by exposing the cancerous cells in a repeated way with shorter intervals without allowing the emergence of resistant clones and by allowing an increase in the intensity of amount. This mode of administration appeared at the same time effective and tolerated very well among patients of more than 70 years. The weekly association of carboplatin and paclitaxel was tested in phase II and showed a rate of response of 14% and one survival 1 year from 31% a randomized test (not dedicated to the old person) of phase II to 3 arms was led by Belani et al.. The best combination of carboplatine + paclitaxel weekly proved to be that associating paclitaxel 100mg/m² 3 weeks out of 4 and carboplatine AUC 6 in J1 with J1 = J29. A test of phase II dedicated the 70 years old to patients and more was carried out in France taking again this association carboplatine (AUC 6) every 4 weeks and paclitaxel weekly (90 mg/m² J1, J8 and J15). This test having included 51 patients highlighted a median of 10,42 months survival (IC 95%: 7,29-17,05)

DETAILED DESCRIPTION:
It thus seemed to us justified to compare a standard arm, the vinorelbine or the gemcitabine (with the choice of the center) in monotherapy with an experimental arm, association carboplatine + paclitaxel. To avoid skewing the results by the introduction of a second line to the choice of the investigator, we chose to force it. It is thus the erlotinib which in a recent test presented by the NCIC at the ASCO 2004 proved its effectiveness in second or third line at the same time in term of response but more especially survival compared to the purely palliative care.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically / cytologically proven NSCLC stage IIIB or IV
* age >= 70 years old and < 90 years old

Ages: 70 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 451 (Actual)
Dates: Start 2006-03; Primary Completion 2010-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1-year

SECONDARY OUTCOMES:
Objective response | 2 cycles

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth QUOIX, Pr, Principal Investigator — Intergroupe Francophone de Cancerologie Thoracique
Locations (5):
- France (5):
  - CH - Pneumologie, Belfort
  - CHU Besancon - Pneumologie, Besançon
  - CHU - Pneumologie, Caen
  - CHU, Grenoble
  - Hôpital Tenon - Pneumologie, Paris

REFERENCES:
- [Background] Pujol JL, Milleron B, Molinier O, Quoix E, Depierre A, Breton JL, Gervais R, Debieuvre D, Hominal S, Namouni F, Tonelli D. Weekly paclitaxel combined with monthly carboplatin in elderly patients with advanced non-small cell lung cancer: a multicenter phase II study. J Thorac Oncol. 2006 May;1(4):328-34. PMID 17409879
- [Result] Quoix E, Zalcman G, Oster JP, Westeel V, Pichon E, Lavole A, Dauba J, Debieuvre D, Souquet PJ, Bigay-Game L, Dansin E, Poudenx M, Molinier O, Vaylet F, Moro-Sibilot D, Herman D, Bennouna J, Tredaniel J, Ducolone A, Lebitasy MP, Baudrin L, Laporte S, Milleron B; Intergroupe Francophone de Cancerologie Thoracique. Carboplatin and weekly paclitaxel doublet chemotherapy compared with monotherapy in elderly patients with advanced non-small-cell lung cancer: IFCT-0501 randomised, phase 3 trial. Lancet. 2011 Sep 17;378(9796):1079-88. doi: 10.1016/S0140-6736(11)60780-0. Epub 2011 Aug 8. PMID 21831418
- [Derived] Quoix E, Westeel V, Moreau L, Pichon E, Lavole A, Dauba J, Debieuvre D, Souquet PJ, Bigay-Game L, Dansin E, Poudenx M, Molinier O, Vaylet F, Moro-Sibilot D, Herman D, Sennelart H, Tredaniel J, Mennecier B, Morin F, Baudrin L, Milleron B, Zalcman G; Intergroupe Francophone de Cancerologie Thoracique. Second-line therapy in elderly patients with advanced nonsmall cell lung cancer. Eur Respir J. 2014 Jan;43(1):240-9. doi: 10.1183/09031936.00048213. Epub 2013 Oct 10. PMID 24114964
- See also: IFCT website — http://www.ifct.fr